CLINICAL TRIAL: NCT03718429
Title: Pharmacodynamic Effects of Low-dose Rivaroxaban in Combination With Antiplatelet Therapies in Patients With Coronary and Peripheral Artery Disease Manifestations
Brief Title: Pharmacodynamic Effects of Low-dose Rivaroxaban With Antiplatelet Therapies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-RIVA01; 20180155 (Other: WIRB)
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Peripheral Arterial Disease; Atrial Fibrillation
Keywords: aspirin; clopidogrel; ticagrelor; rivaroxaban; pharmacodynamic (PD)
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: The proposed investigation will be a prospective PD (pharmacodynamic) study conducted in cohorts of patients with CAD, PAD, or atrial fibrillation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- aspirin (Experimental): Patients on aspirin 81 mg daily will be treated with adjunctive low-dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy will be suspended for 7-10 days.
  Interventions: Drug: Rivaroxaban 2.5 mg Tablet
- aspirin and clopidogrel (Experimental): Patients on aspirin (81 mg daily) plus clopidogrel (75 mg daily) will be treated with adjunctive low-dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy will be suspended for 7-10 days.
  Interventions: Drug: Rivaroxaban 2.5 mg Tablet
- aspirin and ticagrelor (Experimental): Patients on aspirin (81 mg daily) and ticagrelor (90 mg bid) will be treated with adjunctive low-dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy will be suspended for 7-10 days.
  Interventions: Drug: Rivaroxaban 2.5 mg Tablet
- rivaroxaban (No Intervention): A control cohort of subjects with atrial fibrillation on full dose rivaroxaban (20 mg daily) as per standard of care will be recruited and will undergo a single PD assessment.

INTERVENTIONS:
Drug: Rivaroxaban 2.5 mg Tablet — PD assessments will be conducted at 3 time points: i) baseline (while on standard of care antiplatelet therapy), ii) 7-10 days after adjunctive treatment with low dose rivaroxaban, and iii) 7-10 days after dropping aspirin.
  Other Names: Xarelto
  Arms: aspirin; aspirin and clopidogrel; aspirin and ticagrelor

SUMMARY:
Recent studies indicate that anti-factor-Xa inhibition with low-dose rivaroxaban may have a role in the reduction of ischemic recurrences in patients with atherosclerotic disease manifestations.

To date there is very little data, and not conducted in human subjects, on the interplay between anti-Xa blockade with low-dose rivaroxaban and antiplatelet therapies, and in particular how this affects profiles of platelet reactivity and thrombin generation. Given the potential role for the use of low-dose rivaroxaban for the prevention of ischemic recurrences in patients with atherothrombotic disease manifestations, including coronary artery disease (CAD) and peripheral arterial disease (PAD), the study team proposes a prospective pharmacodynamic (PD) investigation assessing the impact of low-dose rivaroxaban when used in combination with antiplatelet treatment regimens commonly used in clinical practice.

DETAILED DESCRIPTION:
Recent studies indicate that anti-factor-Xa inhibition with low-dose rivaroxaban may have a role in the reduction of ischemic recurrences in patients with atherosclerotic disease manifestations.

However, although the introduction of newer antithrombotic strategies has been associated with a reduction in ischemic recurrences in high-risk patients, these have been consistently associated with an increase in bleeding complications. These have been observed particularly with the combination of an oral anticoagulant agent, including low-dose rivaroxaban, with standard DAPT, also known as "triple therapy". Observations from laboratory and clinical studies suggest that in the presence of effective blockade of other pathways triggering thrombotic complications aspirin may not offer added antithrombotic effects but contribute to the increased bleeding. These observations have set the basis for a large number of clinical outcomes studies evaluating whether dropping aspirin in the presence of more potent and effective blockade of other pathways triggering thrombosis has a better safety profile without a tradeoff in efficacy. Amongst these strategies, the use of low-dose rivaroxaban in adjunct to a P2Y12 inhibitor, also known as dual therapy, has been proposed. This approach may be of potential benefit to reduce atherothrombotic complications in high-risk patients following an acute coronary event. On the other hand, regimens with more modest antithrombotic effects compared with a combination of low-dose rivaroxaban and a P2Y12 receptor inhibitor such as low-dose rivaroxaban alone or in combination with aspirin may be more suitable in more stabilized patients.

To date there is very little data, and not conducted in human subjects, on the interplay between anti-Xa blockade with low-dose rivaroxaban and antiplatelet therapies, and in particular how this affects profiles of platelet reactivity and thrombin generation. Given the potential role for the use of low-dose rivaroxaban for the prevention of ischemic recurrences in patients with atherothrombotic disease manifestations, including coronary artery disease (CAD) and peripheral arterial disease (PAD), the study team proposes a prospective pharmacodynamic (PD) investigation assessing the impact of low-dose rivaroxaban when used in combination with antiplatelet treatment regimens commonly used in clinical practice.

ELIGIBILITY:
Inclusion criteria:

* Known CAD (defined as angiographic evidence of >50% coronary artery stenosis or prior coronary revascularization) or PAD (defined as a positive ankle brachial index (ABI) or prior revascularization)
* on treatment with either aspirin (81mg/qd), aspirin (81mg/qd) plus clopidogrel (75mg/qd), or aspirin (81mg/qd) plus ticagrelor (90mg/bid) for at least 3 months per standard of care OR
* Atrial fibrillation (paroxysmal, persistent or permanent) on treatment with rivaroxaban 20 mg qd (if creatinine clearance [CrCl] >50 mL/min) or 15 mg qd (if CrCl 15 - 50 mL/min) per standard of care. Patients with concomitant CAD or PAD who are also taking antiplatelet medications are not eligible. However, if these are only on oral anticoagulation with rivaroxaban (and no antiplatelet therapy) the person will be eligible.

Exclusion criteria:

* Active pathological bleeding, history of clinically significant bleeding events, or deemed at increased risk of bleeding.
* CrCL <20 mL/min
* Any clinical indication to be on triple antithrombotic therapy (DAPT plus an oral anticoagulant)
* An acute coronary event in the past 90 days
* Prior hemorrhagic stroke or intracranial hemorrhage
* Ischemic stroke/transient ischemic attack in the past 6 months
* Chronic use of nonsteroidal anti-inflammatory drugs
* On treatment with combined P-gp and strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, lopinavir/ritonavir, ritonavir, indinavir/ritonavir, and conivaptan) or inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort).
* Known moderate or severe hepatic impairment (Child-Pugh B and C)
* Prior hypersensitivity reaction to rivaroxaban
* On treatment with prasugrel in the past 10 days.
* Platelet count <80x106/mL
* Hemoglobin <10g/dL
* Hemodynamic instability
* Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD,PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Cardiovascular Research Center,, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No
No sharing is planned

REFERENCES:
- [Derived] Galli M, Franchi F, Rollini F, Been L, Jaoude PA, Rivas A, Zhou X, Jia S, Maaliki N, Lee CH, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Geisler T, Jennings LK, Bass TA, Angiolillo DJ. Platelet P2Y12 inhibiting therapy in adjunct to vascular dose of rivaroxaban or aspirin: a pharmacodynamic study of dual pathway inhibition vs. dual antiplatelet therapy. Eur Heart J Cardiovasc Pharmacother. 2022 Sep 29;8(7):728-737. doi: 10.1093/ehjcvp/pvac022. PMID 35353154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 14, 2019 and August 30, 2020 a total of 86 patients were consented for the study.
Pre-assignment Details: 1 patient withdrew the consent before initiation of the study and 3 patients were not eligible to start the study due to the presence of an exclusion criteria.
Groups:
- Aspirin: The cohort of patients on aspirin (81 mg daily) was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Aspirin Plus Clopidogrel: The cohort of patients on aspirin (81 mg daily) plus clopidogrel (75 mg dailiy) was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Aspirin Plus Ticagrelor: The cohort of patients on aspirin (81 mg daily) plus ticagrelor (90 mg bid) was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Rivaroxaban 20 mg: The cohort of patients on rivaroxaban remained on rivaroxaban 20 mg daily.
Period: Baseline Treatment
Arm/Group | Aspirin | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Rivaroxaban 20 mg
Started | 20 | 21 | 21 | 20
Completed | 20 | 21 | 21 | 20
Not Completed | 0 | 0 | 0 | 0
Period: Adjunctive Rivaroxaban 2.5 mg
Arm/Group | Aspirin | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Rivaroxaban 20 mg
Started | 20 | 21 | 21 | 0
Completed | 20 | 20 | 20 | 0
Not Completed | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Period: Stopping Aspirin
Arm/Group | Aspirin | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Rivaroxaban 20 mg
Started | 20 | 20 | 20 | 0
Completed | 20 | 20 | 20 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for each one of the initial 4 treatment cohorts. These already includes patients in other treatment arms were rivaroxaban 2.5 mg was added and aspirin stopped in each patient of each cohort.
Groups:
- Aspirin: The cohort of patients on aspirin was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Aspirin Plus Clopidogrel: The cohort of patients on aspirin plus clopidogrel was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Aspirin Plus Ticagrelor: The cohort of patients on aspirin plus ticagrelor was treated with adjunctive vascular dose rivaroxaban (2.5 mg/bid) for 7-10 days, after which aspirin therapy was suspended for 7-10 days.
- Total: Total of all reporting groups
Arm/Group | Aspirin | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Rivaroxaban 20 mg | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 64 (9) | 59 (9) | 67 (10) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 4 | 9 | 28
  Male | 11 | 14 | 16 | 11 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 12 | 12 | 4 | 36
  White | 11 | 7 | 8 | 16 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
peripheral arterial disease [Count of Participants; unit: Participants] | 4 | 12 | 1 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Platelet-Mediated Global Thrombogenicity
Description: Comparison of platelet-mediated global thrombogenicity measured by light transmittance aggregometry following collagen-related peptide+adenosine diphosphate+ tissue factor (CATF) stimuli between aspirin plus clopidogrel vs. aspirin plus clopidogrel plus rivaroxaban. This was reported as maximal aggregation %. The combination of agonists included in the CATF cocktail leads to activation of multiple platelet pathways including thrombin generation and is therefore a marker of thrombus formation mediated by platelets.
Time Frame: 20 days
Population: For the purpose of this analysis, assessments were conducted in patients with an antithrombotic treatment regimen that paralleled that of the VOYAGER PAD trial, which included patients on triple therapy (DAPT with aspirin 81mg/qd and clopidogrel 75 mg/qd plus rivaroxaban 2.5 mg/bid) and DPI (aspirin 81 mg/qd plus rivaroxaban 2.5 mg/bid). Comparative PD assessments were also made with patients on standard DAPT (aspirin and clopidogrel). Only patients with complete data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Groups:
- Aspirin Plus Clopidogrel: Cohort of patients on aspirin plus clopidogrel
- Aspirin Plus Clopidogrel Plus Rivaroxaban: Cohort of patients on aspirin, clopidogrel and rivaroxaban
- Clopidogrel Plus Rivaroxaban: Cohort of patients on clopidogrel plus rivaroxaban
- Aspirin: Cohort of patients on aspirin only
- Aspirin Plus Rivaroxaban: Cohort of patients on aspirin plus rivaroxaban
- Rivaroxaban: Cohort of patients on rivaroxaban alone
- Aspirin Plus Ticagrelor: Cohort of patients on aspirin plus ticagrelor
- Aspirin Plus Ticagrelor Plus Rivaroxaban: Cohort of patients on aspirin plus ticagrelor plus rivaroxaban
- Ticagrelor Plus Rivaroxaban: Cohort of patients on ticagrelor plus rivaroxaban
- Rivaroxaban 20 mg: Cohort of patients on rivaroxaban 20 mg
Arm/Group | Aspirin Plus Clopidogrel | Aspirin Plus Clopidogrel Plus Rivaroxaban | Clopidogrel Plus Rivaroxaban | Aspirin | Aspirin Plus Rivaroxaban | Rivaroxaban | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor Plus Rivaroxaban | Ticagrelor Plus Rivaroxaban | Rivaroxaban 20 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
percentage of aggregation | 66 (18) | 59 (19) | 69 (18) | 71 (12) | 63 (21) | 74 (10) | 37 (24) | 32 (25) | 35 (24) | 75 (14)
Statistical Analysis 1: Comparison: Aspirin Plus Clopidogrel vs Aspirin Plus Clopidogrel Plus Rivaroxaban; Test type: Superiority — In line with recommendations for pilot investigations, since there were no preliminary data exploring the pharmacodynamic effects of vascular dose rivaroxaban in addition to antiplatelet therapy, we arbitrarily chose a sample size of 20 patients per treatment cohort; p = 0.275, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Platelet Aggregation Measured by VerifyNow PRU
Description: P2Y12 reaction units (PRU) by VerifyNow of dual antiplatelet therapy vs. dual antiplatelet therapy plus rivaroxaban. VerifyNow is a turbidimetric based optical detection system which measures platelet aggregation induced by ADP as an increase in light transmittance.
Time Frame: 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Clopidogrel Plus Rivaroxaban: Cohort of patients on clopidogrel and rivaroxaban
- Aspirin Plus Rivaroxaban: Cohort of patients on aspirin and rivaroxaban
- Rivaroxaban 20 mg: Cohort of patients on rivaroxaban 20 mg only
Arm/Group | Aspirin Plus Clopidogrel | Aspirin Plus Clopidogrel Plus Rivaroxaban | Clopidogrel Plus Rivaroxaban | Aspirin | Aspirin Plus Rivaroxaban | Rivaroxaban | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor Plus Rivaroxaban | Ticagrelor Plus Rivaroxaban | Rivaroxaban 20 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
PRU | 156 (75) | 139 (72) | 156 (73) | 223 (30) | 217 (36) | 229 (34) | 32 (53) | 29 (57) | 36 (61) | 241 (38)
Statistical Analysis 1: Comparison: Aspirin Plus Clopidogrel vs Aspirin Plus Clopidogrel Plus Rivaroxaban; Test type: Superiority; p = 0.488, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Thrombin Generation
Description: Comparison of thrombin generation, reported as peak thrombin level measured by a thrombin generation assay, between aspirin plus clopidogrel vs. aspirin plus clopidogrel plus rivaroxaban. This is reflective of the amount of thrombin that is generated following stimuli with tissue factor. The theombin generation assay will be carried out using Technothrombin® fluorogenic assay kit.
Time Frame: 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µM
Groups:
- Rivaroxaban: Cohort of patients on rivaroxaban 2.5 mg only
Arm/Group | Aspirin Plus Clopidogrel | Aspirin Plus Clopidogrel Plus Rivaroxaban | Clopidogrel Plus Rivaroxaban | Aspirin | Aspirin Plus Rivaroxaban | Rivaroxaban | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor Plus Rivaroxaban | Ticagrelor Plus Rivaroxaban | Rivaroxaban 20 mg
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 20 | 19 | 20 | 19 | 20 | 19
µM | 235 (57) | 135 (79) | 121 (56) | 248 (77) | 130 (54) | 160 (59) | 263 (66) | 162 (83) | 155 (58) | 103 (85)
Statistical Analysis 1: Comparison: Aspirin Plus Clopidogrel vs Aspirin Plus Clopidogrel Plus Rivaroxaban; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 20 days
Description: During study treatment, ischemic cardiac events (including death, myocardial infarction, stroke, or urgent revascularization) and serious adverse events (bleeding and other adverse events) were collected. Given the low number of adverse events (only 1 event occurred), events are reported per cohort. The single event reported occurred in the aspirin plus clopidogrel plus rivaroxaban treatment group.
Groups:
- Rivaroxaban: The cohort of patients on rivaroxaban remained on rivaroxaban 20 mg daily.
Arm/Group | Aspirin | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=20) | Aspirin Plus Clopidogrel (N=21) | Aspirin Plus Ticagrelor (N=21) | Rivaroxaban (N=20)
Bleeding (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — Minor bleeding defined as Bleeding Academic Research Consortium (BARC) type 2 bleeding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03718429/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT03718429/ICF_001.pdf